CLINICAL TRIAL: NCT03104907
Title: Prostatic Artery Embolization for Obstructive Uropathy Due to Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Brian Malling, MD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-17000714-2
Record Dates: First submitted 2017-03-28; First posted 2017-04-07 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Prostatic Neoplasm; Lower Urinary Tract Symptoms; Urological Manifestations; Prostatic Diseases
Keywords: IPSS; Quality of Life; DAN-PSS; Complications; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Lower Urinary Tract Symptoms; Urological Manifestations; Prostatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostatic Artery Embolization (Experimental): Embolization of the prostatic arteries to induce necrosis and a reduction of the prostate volume.
  Interventions: Procedure: Prostatic Artery Embolization

INTERVENTIONS:
Procedure: Prostatic Artery Embolization — The procedure is performed with the patient under local anaesthetic and if necessary sedation. We will be using a percutaneous transfemoral approach, super-selective catheterisation of small prostatic arteries is carried out using microcatheters. Embolisation will be done using microspherical embolic material.

SUMMARY:
The aim of this study is to investigate the safety and efficacy of prostatic artery embolization of patients with recurrent symptoms secondary to locally advanced prostatic cancer including pelvic pain, bleeding or need for permanent urinary catheter who are unfit for or refuse surgical treatment.

DETAILED DESCRIPTION:
This is a prospective study investigating the safety and efficacy of PAE for patients with prostate cancer who suffers from acute urinary retention, severe LUTS and/or recurrent complications such as haematuria.

Our hypothesis is that PAE will eliminate the need for indwelling catheter and improve IPSS and QoL 12 months post-procedure.

1, and 6 months follow-up.

Main outcome Ability to void after removal of indwelling catheter

Secondary outcomes International Prostate Symptom Score (IPSS) Quality of Life (QoL) International Index of Erectile Function (IIEF) Prostate volume Peak void flow (Qmax) Post-void residual (PVR) Classify complications according to Society of Interventional Radiology (SIR) guidelines for reporting Prostate-specific antigen (PSA)

ELIGIBILITY:
Inclusion Criteria:

* Indwelling catheter secondary to locally advanced prostate cancer (PCa) or
* Moderate-severe Obstructive LUTS secondary to PCa
* Unsuitable for or refuse surgery

Exclusion Criteria:

* Bladder dysfunction(and known neurological conditions affecting bladder function)
* Urethral strictures
* Bladder neck contracture
* Known sphincter anomalies
* Big bladder diverticulum or stones
* Kidney insufficiency (eGFR < 45)
* Coagulation disturbances
* Severe atheromatous or tortuosity of arteries
* Allergy to contrast medium
* Unable to undergo MR imaging
* Bladder malignancy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Ability to void spontaneously | 1 months
  The ability to void after removal of the indwelling catheter

SECONDARY OUTCOMES:
IPSS | 1, 6 months
  International Prostate Symptom Score
QoL | 1, 6 months
  Quality of Life (scale)
IIEF | 1, 6 months
  International Index of Erectile Function
PV | 1, 6 months
  Prostate Volume
PVR | 1, 6 months
  Post-void residual
Qmax | 1, 6 months
  Peak void flow
PSA | 1, 24-hours, 6 months
  Prostate-specific antigen

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lönn, Professor, Study Chair — Radiologisk Klinik, Rigshospitalet
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malling B, Roder MA, Lindh M, Frevert S, Brasso K, Lonn L. Palliative Prostate Artery Embolization for Prostate Cancer: A Case Series. Cardiovasc Intervent Radiol. 2019 Oct;42(10):1405-1412. doi: 10.1007/s00270-019-02227-4. Epub 2019 May 6. PMID 31062066